CLINICAL TRIAL: NCT05833581
Title: Examining the Reliability and Validity of the New York Heart Association Classification Guide to Assign Class for Patients With Heart Failure and Application Into Practice
Brief Title: Consistently Assess Signs and Symptom of Heart Failure
Acronym: CLASS-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Board of Trustees of Illinois State University (Other)
Collaborators: University of Colorado, Denver (Other); Lancaster General Hospital (Other); University of North Carolina, Greensboro (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Marilyn Prasun, Professor, Carle BroMenn Medical Center Endowed Professor, Board of Trustees of Illinois State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HF-2021-000136
Record Dates: First submitted 2023-03-28; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A prospective cross-sectional study in the ambulatory care settings that manages adult patients with chronic heart failure (both heart failure with reduced ejection fraction [HFrEF] and heart failure with preserved ejection fraction [HFpEF]).
Masking Description: For the 6-minute walk test the technician performing the test is masked. The remainder of the data is not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Intervention Study Arm (Experimental): All participants with HF will be evaluated by their HF providers who will use the NYHA Classification Guide to assist with assignment of HF class. The participant will then complete a 6-minute walk test. Subsequently participating providers will utilize the guide to assess and assign the class of their HF patients in practice.
  Interventions: Other: New York Heart Association Classification Guide

INTERVENTIONS:
Other: New York Heart Association Classification Guide — The New York Heart Association Classification Guide is a questionnaire that assists in guiding the provider in selection of the patient's class

SUMMARY:
Heart failure (HF) is a major public health problem. The New York Heart Association (NYHA) Functional Classification by a HF provider helps to guide their decisions in patient treatment. The purpose of this study is to further examine the NYHA Classification Guide that is designed to assist healthcare providers. The investigators will conduct the study in the outpatient clinic setting where adult patients with chronic heart failure are treated. HF providers will be asked to complete the NYHA classification Guide and then participants will complete a standardized 6-minute walk test which is considered as the gold standard. Participant results will be compared between providers' assigned class and the results from the 6-minute walk test. The subsequent phase of the study will be incorporation of the NYHA Classification Guide into clinical practice. HF providers will use the NYHA Classification Guide for 30 days in the clinic setting and will report their perceptions.

DETAILED DESCRIPTION:
As a continuation of prior work, the purpose of this study is to further examine the reliability and validity of the New York Heart Association (NYHA) Classification Guide and application into practice. The investigators will conduct a prospective cross-sectional study in the ambulatory care settings that manages adult patients with chronic heart failure (both heart failure with reduced ejection fraction [HFrEF] and heart failure with preserved ejection fraction [HFpEF]). HF providers will be asked to complete the NYHA classification Guide and assign one of 4 functional classes: Class I, Class II, Class III, or Class IV. Participants will then complete a standardized 6-minute walk test (6MWT), considered as the gold standard. Participant results will be compared between providers' assigned class and the results from the 6-minute walk test. The subsequent phase of the study will be incorporation of the NYHA Classification Guide into clinical practice. Clinicians will utilize the NYHA Classification Guide for 30 days and will report perceived barriers and facilitators. Data reporting NYHA Class and HF Stage will be obtained from 30 days prior implementation and compared to during implementation.

ELIGIBILITY:
Participant Inclusion Criteria:

* A documented confirmed diagnosis of Heart Failure (HF)
* Under the care of a Cardiologist and/or Advanced Practice Provider working in Cardiology
* 18 years of age or older and less than 90 years of age
* Alert and oriented to person, place, and time
* Ability to walk without assistance
* Able to read and speak English

Participant Exclusion Criteria:

* Diagnosed with myocardial infarction, coronary artery bypass graft (CABG), angioplasty or stent in the previous 30-days
* Unstable angina in the previous 30 days
* Active endocarditis
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled hypertension with systolic blood pressure readings > 180 mmHg or diastolic pressure readings > 100 mmHg
* Uncontrolled atrial dysrhythmia or 3rd degree heart block
* Active ventricular arrhythmias resulting in 1 or more shocks in the past month
* Acute pulmonary embolus or pulmonary infection
* Thrombosis of the lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Room air oxygen saturation (SPO2) at rest less than 90%
* Acute respiratory failure
* Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise such as, infection, thyrotoxicosis
* Left ventricular assist device
* Mental impairment leading to inability to cooperate

Provider Inclusion Criteria:

• Licensed healthcare providers (Physicians and Advance Practice Providers) in HF ambulatory clinical sites who care for adult patients with HF.

Providers Exclusion Criteria:

• Providers who do not actively manage adult patients with HF.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-12-17 (Estimated); Study Completion 2024-06-17 (Estimated)

PRIMARY OUTCOMES:
Reliability of the New York Heart Association (NYHA) Classification Guide | 12 weeks
  Experts will assign NYHA class using the guide in 30 selected clinical records. The assigned class results will be compared to determine reliability.
Validity of the New York Heart Association (NYHA) Classification Guide | 1 year
  Providers will assign NYHA class using the guide to assess participants with HF who will then perform a 6-minute walk test.
Barriers to implementation of the New York Heart Association (NYHA) Classification Guide | 30-days
  Providers will be surveyed following 30-days of using the NYHA Classification Guide in the clinical setting regarding perceived barriers to implementation into practice.
Facilitators to implementation of the New York Heart Association (NYHA) Classification Guide | 30-days
  Providers will be surveyed following 30-days of using the NYHA Classification Guide in the clinical setting regarding perceived facilitators to implementation into practice.
Documentation after Implementation of the New York Heart Association (NYHA) Classification Guide | 60-days
  30-days prior and 30-days during implementation of the NYHA Classification Guide in clinical practice, the provider clinic notes from the patient visit will be assessed for documentation of NYHA class (I-IV) and HF stage (A-D).

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn A. Prasun, PhD, Principal Investigator — Board of Trustees of Illinois State University
Locations (3):
- United States (3):
  - University of Colorado Medical Center, Aurora, Colorado
  - Carle BroMenn Medical Center, Normal, Illinois
  - Lancaster General Health/Penn Medicine, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be published.

REFERENCES:
- See also: Providers' Accuracy in Decision-Making with Assessing NYHA Functional Class of Patients with Heart Failure after use of a Classification Guide — http://doi.org/10.1016/j.hrtlng.2022.03.017
- See also: Providers' assignment of NYHA functional class in patients with heart failure: A vignette study — http://doi.org/10.1016/j.hrtlng.2021.07.009